CLINICAL TRIAL: NCT04578964
Title: Determining the Cardiovascular Risk Factors Affecting the Age of First Acute Coronary Syndromes
Brief Title: Determining the Age of First Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz Demirci, principal investigator, Antalya Training and Research Hospital
Other Study IDs: 2014-097
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Acute Coronary Syndrome; Age Problem; Risk Factor, Cardiovascular
Keywords: acute coronary syndrome; age; obesity; risk factor, Cardiovascular; smoking; gender; hyperlipidemia; diabetes mellitus; psychosocial stress
MeSH Terms: conditions — Acute Coronary Syndrome; Obesity; Smoking; Coitus; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to evaluate the association between the obesity grade and the age of the first acute coronary syndrome (ACS). The effect of cardiovascular (CV) risk factors and the age of first ACS in patients with severe obesity was also examined. Consecutive patients with diagnosis of first episode of ACS were prospectively enrolled in 2014 to 2024.Cardiovascular risks of patients will be determined according to clinical and laboratory evaluation and patients were categorized by their body mass indices (BMI). Independent variables that effected the age of first ACS were examined by linear regression analysis

DETAILED DESCRIPTION:
In the first stage, the first ACS diagnosis of the patients will be tried to be clarified. It will be tried to clarify whether the patients have had ACS before, according to their history, ecg echo and coronary angiography findings. Patients with previous ACS or uncertain ACS diagnosis will not be included in the study.

In the second stage, cardiovascular risk burdens of patients for whom the initial ACS diagnosis is clear will be revealed. Smoking, diabetes mellitus (DM), hypertension (HT), psychological stress, socio-economic status, migration history, cholesterol parameters will be determined. The duration and severity of these risk factors will be determined. In the final model, each risk factor will be examined in detail with its sub-tabs and the effect of each risk factor will be examined separately.

Eventually, a model will be developed that allows predicting the first ACS age. The shortcomings of this model and the narrow scope of the definition of the population will be determined and the direction will be determined for the studies that improve these points.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with the diagnosis of the first acute coronary syndrome

Exclusion Criteria:

* Previous cardiovascular disease
* Chronic renal disease,
* Chronic obstructive pulmonary disease,
* Malignancy,
* Regularly use of statins, antiplatelets or anticoagulants,
* Situations where oral communication cannot be established with the patient
* Situations when coronary angiography (CAG) could not be performed .
* Patients with findings that might be related to previous MI on electrocardiography (ECG) or echocardiography and total occlusion other than 'culprit' lesion and no critical stenosis on CAG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First acute coronary syndrome patients admitted to the coronary intensive care unit
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-02 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Determining the effect of cardiovascular risk factors on the mean age of the first acute coronary syndrome | 10 years
  Detection of the effect of gender, smoking, obesity, diabetes, hypertension, psychological stress, socioeconomic status, migration, dyslipidemia on the age of first acute coronary syndrome episode.

SECONDARY OUTCOMES:
Determining the effect of obesity on the mean age of the first acute coronary syndrome | 6 years
  Grouping will be made to obesity degree (Normal, overweight, obesity severe obesity). The first ACS average age of these groups will be compared. Risk factors affecting this average age will not be revealed by linear regression model.
Determining the effect of migration on the mean age of the first acute coronary syndrome. | 6 years
  Do the patients live in the city where they were born. It will be determined whether he migrated from another city. If there is a migration situation, the reasons will be determined. The migration direction will be determined according to the regions. The impact of migration and migration direction on the first ACS age will be determined.
Model for calculating the acute coronary syndrome age | 8 years
  Develop a model that calculates the estimated age of ACS on the basis of cardiovascular risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Deniz Demirci, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Demirci D, Demirci DE, Chi G. Association between obesity grade and the age of the first acute coronary syndrome: Prospective observational study. Int J Cardiol. 2022 Mar 15;351:93-99. doi: 10.1016/j.ijcard.2021.11.080. Epub 2021 Dec 2. PMID 34864079